CLINICAL TRIAL: NCT05160090
Title: Single Dose Crossover Comparative Bioavailability Study of Bupropion Hydrochloride Modified Release Tablet 300mg In Healthy Adult Subjects / Fasting State
Brief Title: Single Dose Crossover Comparative Bioavailability Study of Bupropion Hcl MR Tablet 300mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alembic Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: AMC-P7-739
Record Dates: First submitted 2021-11-22; First posted 2021-12-16 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Bioequivalence
MeSH Terms: interventions — Bupropion

STUDY DESIGN:
Intervention Model Description: Single center, randomized, single dose, laboratory-blinded, 2-period, 2-sequence, crossover design
Masking Description: Open label (laboratory blind)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test- BUPROPION HCl MR TABLETS 300mg (Active Comparator): Single dose of Test- BUPROPION HCl MR TABLETS 300mg
  Interventions: Drug: Bupropion HCl MR tablets 300mg
- Reference-Elontril 300 mg (Active Comparator): Elontril 300 mg (Bupropion HCl MR tablets 300mg)
  Interventions: Drug: Bupropion HCl MR tablets 300mg

INTERVENTIONS:
Drug: Bupropion HCl MR tablets 300mg — In each study period, a single 300 mg dose of Bupropion will be administered orally with about 240 mL of water at ambient temperature, in the morning, while subjects are seated, following a 10-hour overnight fast.
  Other Names: Reference-Elontril (Bupropion HCl) MR tablets 300mg

SUMMARY:
The objective of this study is to determine the bioequivalence of 2 different formulations of bupropion after a single oral dose administration under fasting conditions.

The secondary objective of this study is to evaluate the safety and tolerability of the Test and Reference formulations in healthy subjects.

DETAILED DESCRIPTION:
This is a single center, randomized, 2-treatment, 2-period, 2-sequence, crossover, single dose study design, in which 34 healthy adult subjects will receive 1 of the study treatments during each study period.

Subject eligibility for this study will be determined at the screening visit and eligible subjects will be admitted to the clinical research unit at least 10 hours prior to drug administration for each study period.

For each study period, subjects will receive a single 300 mg oral dose of bupropion, under fasting conditions and undergo a 96-hour PK sample collection. Subjects are to be discharged from the clinic after the 36-hour postdose PK sample collection, and following medical approval. However, they may be advised to stay at the clinical site for safety reasons, if judged necessary by the physician in charge. Subjects will return to the clinic for blood collections at 48, 72, and 96 hours postdose.

The drug administrations in each period will be separated by at least 14 calendar days.

The duration of the clinical portion of this study (excluding the screening period) is expected to be approximately 19 days. The actual overall study duration may vary.

Tests during study:

An alcohol breath test will be performed before each period of the study. Screening for drugs of abuse will be performed before each period of the study. A C-SSRS questionnaire will be performed prior to each study period, as well as before discharge of each period. Neurologic Function Test will be performed at screening, approximately 26 hours after each drug administration & end of the study.

For female subjects, a serum pregnancy test will be performed before each period of the study & end of study.

Vital signs will be measured prior to and approximately 2.5, 4, 6, 12, 24, and 36 hours following each drug administration.

Safety assessments will include physical examination, vital signs, clinical laboratory tests, neurologic function tests, and AE monitoring. Additional safety measurements may be performed at the discretion of the investigator for reasons related to subject safety.

The physician in charge will be present at the clinical site for at least the first 6 hours following each drug administration and will remain available at all times throughout the study.

Post study Tests:

Hematology, general biochemistry (including a serum pregnancy test for female subjects), and urinalysis tests will be repeated along with the collection of the last blood sample of the study.

A complete physical examination (including vital signs) will also be performed.

Bioanalysis: Bupropion & its metabolites plasma concentrations will be measured by a validated bioanalytical method.

Standards for Bioequivalence:

Statistical inference of bupropion will be based on a bioequivalence approach using the following standards:

The ratio of geometric LSmeans with corresponding 90% confidence interval calculated from the exponential of the difference between the Test and Reference products for the ln-transformed parameters Cmax, AUC0-T, AUC0-∞, should all be within the 80.00 to 125.00% bioequivalence range.

For the metabolites (hydroxybupropion, threohydrobupropion and erythrohydrobupropion) , the same criteria will be applied and the results will be presented as supportive evidence of comparable therapeutic outcome.

ELIGIBILITY:
Inclusion Criteria

1. Provision of signed and dated informed consent form (ICF)
2. Subjects able to communicate effectively with study personnel
3. Stated willingness to comply with all study procedures and availability for the duration of the study
4. Healthy adult male or female
5. If female, meets 1 of the following criteria

   1. Is of childbearing potential and agrees to use an acceptable contraceptive method. Acceptable contraceptive methods include Abstinence from heterosexual intercourse from at least 28 days prior to the first study drug administration through to at least 30 days after the last dose of the study drug

      1 of the following highly-effective contraceptive methods, used from at least 28 days prior to the first study drug administration through to at least 30 days after the last dose of the study drug Intrauterine device (without hormones) Male partner vasectomized at least 6 months prior to the first study drug administration Male condom with spermicide In addition of the male condom with spermicide, female needs to use an additional method from the first study drug administration through to at least 30 days after the last dose of the study drug Diaphragm/cervical cap Or
   2. Male partner has had a vasectomy less than 6 months prior to dosing, and agrees to use an additional acceptable contraceptive method from the first study drug administration through to at least 30 days after the last dose of the study drug Or
   3. Is of non-childbearing potential, defined as surgically sterile (i.e. has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation) or is in a postmenopausal state (i.e. at least 1 year without menses without an alternative medical condition prior to the first study drug administration)
6. Aged at least 18 years but not older than 45 years
7. Body mass index (BMI) greater than or equal to 18.50 kg/m2 and below 30.00 kg/m2
8. Minimal body weight of 60 kg
9. Non- or ex-smoker (An ex-smoker is defined as someone who completely stopped using nicotine products for at least 180 days prior to the first study drug administration)
10. Clinical laboratory values within the laboratory's stated normal range; if not within this range, they must be without clinical significance, as determined by an investigator
11. Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on the physical examination (including vital signs) and/or electrocardiogram (ECG), as determined by an investigator

Exclusion Criteria

1. Female who is lactating at screening
2. Female who is pregnant according to the pregnancy test at screening or prior to the first study drug administration
3. Difficulty with donating blood due to bad veins
4. Difficulty in swallowing tablets or capsules
5. Seated blood pressure lower than 100/60 mmHg at the screening visit and prior to the first study drug administration
6. History of significant hypersensitivity to bupropion or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
7. Presence or history of significant gastrointestinal, liver or kidney disease, or any other condition that is known to interfere with drug absorption, distribution, metabolism or excretion, or known to potentiate or predispose to undesired effects
8. History of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease
9. Showing suicidal tendency as per the Columbia Suicide Severity Rating Scale (C-SSRS) administered at screening (APPENDIX 6 COLUMBIA-SUICIDE SEVERITY RATING SCALE (C-SSRS) BASELINE/SCREENINGVERSION)
10. Presence of out-of-range cardiac interval (PR < 110 msec, PR > 200 msec, QRS < 60 msec, QRS >110 msec and QTcF > 440 msec) on the ECG at screening or other clinically significant ECG abnormalities, unless deemed non-significant by an investigator
11. Use of concomitant medications that lower seizure threshold, including but not limited to: antipsychotics, antidepressants, lithium, amantadine, theophylline, systemic steroids, quinolone antibiotics, and anti-malarials
12. Use of over-the-counter stimulants or anorectics
13. Maintenance therapy with any drug or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
14. Any clinically significant illness in the 28 days prior to the first study drug administration
15. Use of any prescription drugs in the 28 days prior to the first study drug administration, that in the opinion of an investigator would put into question the status of the participant as healthy
16. Any history of tuberculosis
17. Positive test result for alcohol and/or drugs of abuse at screening or prior to the first drug administration
18. Positive screening results to HIV Ag/Ab combo, hepatitis B surface antigen or hepatitis C virus tests
19. Inclusion in a previous group for this clinical study
20. Intake of bupropion in the 28 days prior to the first study drug administration
21. Intake of an Investigational Product (IP) in the 28 days prior to the first study drug administration
22. Intake of an IP in another clinical trial with a long half-life (≥120 hours) in the previous 90 days prior to the first study drug administration
23. Donation of 50 mL or more of blood in the 28 days prior to the first study drug administration
24. Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the 56 days prior to the first study drug administration

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2020-01-18 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
Cmax | Up to 96.00 hours
  Maximum observed concentration occurring at time Tmax
AUC0-T | Up to 96.00 hours
  Area under the concentration time curve from the time of last dosing to Tlast.
AUC0-∞ | Up to 96.00 hours
  Area under the concentration time curve extrapolated to infinity, calculated as AUCT + ĈLQC/λZ, where ĈLQC is the predicted concentration at time Tlast

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sicard, MD, Principal Investigator — Clinical Investigator
Locations (2):
- Canada (2):
  - Algorithme Pharma Inc., Mount Royal, Quebec
  - Algorithme Pharma, Mount Royal, Quebec

IPD SHARING:
Plan to Share IPD: No